CLINICAL TRIAL: NCT04171427
Title: Evaluation of the Efficacy and the Cutaneous Acceptability of a Dermocosmetic Product in the Repigmentation of Vitiligo -Study Realized by a Dermatologist-
Brief Title: Evaluation of the Efficacy and the Cutaneous Acceptability of a Dermocosmetic Product in the Repigmentation of Vitiligo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Laboratoire Dermatologique ACM (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18E1721
Record Dates: First submitted 2019-11-07; First posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-10

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Intervention Model Description: Three parallel groups testing different dosages / combinations of treatments
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lithium liposome and placebo A (Other): • Group A : 4 patients; Lithium liposome 1 application / day (evening) on target lesions on one side of the body, placebo 1 application / day (evening) on contralateral target lesions and excimer lamp on target lesions on the two sides;
  Interventions: Other: Lithium liposome; Other: Placebo
- Lithium liposome and placebo B (Other): Group B : 4 patients; Liposomal Lithium 2 applications / day (morning and evening) on target lesions on one side of the body, placebo 2 applications / day (morning and evening) on contralateral target lesions and excimer lamp on target lesions on the two sides;
  Interventions: Other: Lithium liposome; Other: Placebo
- Lithium liposome and placebo C (Other): Groupe C : 4 patients; Lithium liposome 2 applications / day (morning and evening) on one side, placebo 2 applications / day (morning and evening) on contralateral target lesions.
  Interventions: Other: Lithium liposome; Other: Placebo

INTERVENTIONS:
Other: Lithium liposome — Cosmetic product
Other: Placebo — Cosmetic product vehicle

SUMMARY:
* Study in proof of concept;
* Double blind study;
* Comparative study, versus placebo in intra-individual
* Three parallel groups testing different dosages / combinations of treatments
* Randomized.

DETAILED DESCRIPTION:
This study has as objectives:

Primary objective :

• Evaluate the percentage of repigmentation observed one month after the end of three months of treatment measured on an objective layer by image analysis;

Secondary objectives:

Evaluate:

* the percentage of repigmentation observed after one, two and three months of treatment measured on an objective layer by image analysis;
* the ability of the product to maintain the human body in good condition (cutaneous acceptability) by clinical examination by the dermatologist;
* Patient satisfaction using a visual analogue scale from 0 to 10.
* The illustrative effect using standardized photographs;
* The quantity of product by weighing the tubes.
* The occurrence of possible adverse effects.

Population:

* Sexe: female and male;
* Age: over 18 years old;
* Patients with stable non-segmental vitiligo lesions (defined as no new lesions or lesions that have been present for at least 3 months, lack of hypochromic margins in Wood's lumen and absence of confetti depigmentation);
* Patients with 2 to 6 symmetrical lesions (1 to 3 on each side). These lesions (macules) will be treated for a minimum surface of 2 cm² and a maximum surface of 100 cm².

ELIGIBILITY:
•Inclusion Criteria: Sexe: female and male;

* Age: over 18 years old;
* Patients with stable non-segmental vitiligo lesions (defined as no new lesions or lesions that have been present for at least 3 months, lack of hypochromic margins in Wood's lumen and absence of confetti depigmentation);
* Patients with 2 to 6 symmetrical lesions (1 to 3 on each side). These lesions (macules) will be treated for a minimum surface of 2 cm² and a maximum surface of 100 cm².
* Healthy volunteer;
* Volunteer having given in writing his free, informed and express consent;
* Volunteer willing to abide by the protocol and procedures of the study.

Exclusion Criteria:

* Pregnant woman or woman who is breastfeeding or planning for early pregnancy during the study;
* Patient with segmental or mixed vitiligo;
* Patient with vitiligo of the external genitalia;
* Patient with vitiligo touching hands and feet only
* Patient with a history of skin cancer or pre-cancerous skin lesions;
* Patient taking topical or systemic vitiligo treatments in the month prior to the start of the study;
* Patient taking concomitant local or general corticosteroid therapy or immunomodulatory therapy;
* Patient with a history of photodermatoses or taking photosensitizing medications;
* Patient having planned to expose himself (artificial sun or UV) during the study at the level of the zones to be treated and / or having been exposed during the month preceding the beginning of the study and having an acquired pigmentation (tanning) obvious;
* Patient who had been treated with phototherapy within 4 weeks before randomization;
* Patient with lithium allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-11-21 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
the percentage of repigmentation | 4 months
  • Evaluate the percentage of repigmentation observed one month after the end of three months of treatment measured on an objective layer by image analysis;

SECONDARY OUTCOMES:
the percentage of repigmentation and acceptability | 1 month, 2 months, 3 months
  the percentage of repigmentation observed after one, two and three months of treatment measured on an objective layer by image analysis;
  * the ability of the product to maintain the human body in good condition (cutaneous acceptability) by clinical examination by the dermatologist;
  * Patient satisfaction using a visual analogue scale from 0 to 10.
  * The illustrative effect using standardized photographs;
  * The quantity of product by weighing the tubes.
  * The occurrence of possible adverse effects.

CONTACTS AND LOCATIONS:
Overall Officials: Samy FENNICHE, Principal Investigator — Hbib Thamer Hosptal
Locations (1):
- Hbib thamer Hospital, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-25): https://cdn.clinicaltrials.gov/large-docs/27/NCT04171427/Prot_SAP_000.pdf